CLINICAL TRIAL: NCT02901054
Title: Investigation of Cerebrospinal Fluid (CSF) Pharmacokinetics of Ondansetron
Brief Title: CSF Pharmacokinetics of Ondansetron
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, simon.haroutounian, Assistant Professor, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201605080
Record Dates: First submitted 2016-09-04; First posted 2016-09-15 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label infusion ondansetron (Experimental): 1. A single 4-mL CSF sample per subject.
  2. Serial blood sampling at 0 (pre-infusion), 15, 30, 60, 120, and 180 min after ondansetron administration
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — A single 15-min intravenous infusion of ondansetron
  Other Names: Zofran

SUMMARY:
Serotonergic 5-HT3 receptors in the central nervous system are involved in pain processing after nerve injury. We are interested in learning if 5-HT3 receptor antagonist ondansetron might be an appropriate drug for treating pain after nerve injury (neuropathic pain), by investigating its bio-distribution in the cerebro-spinal fluid, and the genetic variability that may affect that distribution.

Study procedures will include iv ondansetron administration, serial blood draws, cerebrospinal fluid (CSF) sampling, pregnancy testing, and possible ECG.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years old;
2. Patients planned to undergo hip or knee arthroplasty with spinal anesthesia;
3. Ability to provide informed consent

Exclusion Criteria:

1. Not giving consent to participate in the study;
2. Patients with history of or current hepatic or renal insufficiency;
3. Patients with BMI ≥ 33;
4. Patients with heart failure or active arrhythmias;
5. Patients with severe systemic disease that is a constant threat to life;
6. Contraindication or allergy to ondansetron;
7. Pregnancy or lactation.
8. Prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2016-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Dept of Anesthesiology, Washington Univ School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 consented, 3 participants withdrew prior to any intervention, and 1 participant excluded before outcomes data collection
Groups:
- Open Label Infusion Ondansetron: The full study cohort (open label, no treatment allocation)
Period: Overall Study
Arm/Group | Open Label Infusion Ondansetron
Started | 19 (19 consented, 3 withdrew prior to intervention, 1 received study drug but surgery was cancelled.)
Completed | 15
Not Completed | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Open Label Infusion Ondansetron: The entire cohort of subjects in this open-label study
Arm/Group | Open Label Infusion Ondansetron
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: one subject withdrew due to cancelled surgery. data not analyzed
  Participants
    number analyzed (Participants) | 15
    Female | 8
    Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: one subject withdrew due to cancelled surgery. data not analyzed
  Participants
    number analyzed (Participants) | 15
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 14
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Washington University Population: One subject withdrew due to cancelled surgery. Data were not analyzed.
  participants
    United States: number analyzed (Participants) | 15
    United States | 15

OUTCOME MEASURES:

1. Primary Outcome: CSF to Plasma Concentration Ratio
Description: CSF: plasma ratio of ondansetron at the time of obtaining the CSF sample
Time Frame: 0-180 min from the beginning of infusion
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Open Label Infusion Ondansetron
Number analyzed (Participants) | 15
Ratio | 0.15 (0.05)

ADVERSE EVENTS:
Time Frame: During the infusion of the study drug and up to the surgery start (1 day)
Groups:
- Open Label Infusion Ondansetron: The entire cohort of patients in this open-label study
Arm/Group | Open Label Infusion Ondansetron
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT02901054/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT02901054/Prot_SAP_001.pdf